CLINICAL TRIAL: NCT07076849
Title: Mechanistic Pathways of Probiotic Supplementation in Optimizing Iron and Hematological Status Among Pregnant Females at Risk of Iron Deficiency Anemia
Brief Title: Probiotic Supplementation in Optimizing Iron and Hematological Status Among Pregnant Females
Acronym: ProMoms
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-0431
Record Dates: First submitted 2025-07-09; First posted 2025-07-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-01

CONDITIONS: Iron Deficiency (ID); Pregnancy
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactiplantibacillus plantarum 299v (LP299V®) (Experimental): Probiotic
  Interventions: Dietary Supplement: Lactiplantibacillus plantarum 299v
- Control (Placebo Comparator): Placebo capsule
  Interventions: Other: Placebo Capsule(s)

INTERVENTIONS:
Dietary Supplement: Lactiplantibacillus plantarum 299v — Probiotic
  Arms: Lactiplantibacillus plantarum 299v (LP299V®)
Other: Placebo Capsule(s) — Placebo control
  Arms: Control

SUMMARY:
Maternal iron deficiency (ID) and iron deficiency anemia (IDA) is associated with maternal and infant mortality, spontaneous preterm birth, maternal postpartum hemorrhage, and neurocognitive defects in the neonate. Therefore, preventing maternal IDA in at-risk women is critical. The standard approach to improving iron status in pregnancy (i.e., oral iron supplements) is suboptimal and gastrointestinal discomforts associated with this approach (i.e., constipation) impairs adherence. The incidence of ID (18%) and IDA (5%) in pregnant populations suggest alternative interventions are needed to optimize iron status in pregnancy. There is increasing evidence that consuming the probiotic Lactoplantibacillus plantarum 299v (LP299V®) can enhance dietary non-heme iron absorption by changes in the composition and metabolic patterns of gut microbiota that reduce intestinal pH, enhance mucin production and favor an anti-inflammatory milieu. This immunomodulatory effect may be important because inflammation stimulates hepatic production of hepcidin, a master regulator of systemic iron homeostasis, which inhibits iron flow into circulation from diet and body stores. Further, the effects of LP299V® may extend to the placenta. The investigators' team showed previously that maternal iron deficiency is associated with changes to placental iron metabolism with more iron sequestered in the placenta and less iron transferring to the fetus. Given its positive effects on maternal iron status, the investigators surmise that LP299V® supplementation will result in higher placenta protein expression of iron transporters, transferrin receptor-1 and ferrroportin-1, and lower placental iron accumulation/content. The primary goal of this study is to test the efficacy of this low-cost, safe, innovative approach to optimizing maternal iron status in individuals at risk for ID in pregnancy [Hb 11.0 - 11.9 g/dL (first trimester) and Hb 10.5 - 11.5 g/dL (second trimester) based on new OB clinical complete blood count (CBC) results obtained from the EHR] from 10-16 weeks gestational age (GA) until the time of labor. The investigators will also test the effects on neonatal (cord blood) iron status and (cord blood + newborn heel stick) Hb at birth and determine the effect of maternal LP299V® supplementation on the maternal gut microbiome, hepcidin-ferroportin axis and placenta iron and placenta transport of iron as its primary mechanisms of action. Finally, the investigators will explore the effect of maternal LP299V® supplementation on infant neurodevelopment at birth. This study is an essential first step toward evaluating if twice daily oral LP299V® is an efficacious, safe, inexpensive, and scalable clinical strategy for the prevention of maternal ID and its related complications in at-risk women.

ELIGIBILITY:
Inclusion Criteria:

* singleton naturally conceived pregnancy;
* at risk of IDA [Hb 11.0 - 11.9 g/dL (first trimester) and Hb 10.5 - 11.5 g/dL (second trimester) based on new OB clinical complete blood count (CBC) results obtained from the EHR;
* 18 - 45 years old;
* 10-16 weeks GA;
* fluency in English to provide consent and complete study procedures;
* ability to provide consent;
* and ownership of a smartphone (currently more than 90% of our patient population at the CWH).

Exclusion Criteria:

* IDA or other nutritional anemia (i.e., diagnosed or suspected B12 or folate deficiency) based on new OB blood work that includes MCV and MCH to characterize the anemia;
* recent blood transfusion;
* autoimmune disorder (e.g., rheumatoid arthritis);
* inflammatory bowel disease;
* oral or IV antibiotic use within 2 months;
* previous spontaneous preterm birth;
* history of bariatric surgery;
* malabsorptive disease;
* current hyperemesis;
* current eating disorder;
* hematologic disorder or trait carrier (e.g., hemochromatosis, β-thalassemia);
* current tobacco, alcohol or illicit drug use (Excluding marijuana).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2030-10-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Maternal hemoglobin from complete blood count (CBC) with differential | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw

SECONDARY OUTCOMES:
Maternal iron deficiency anemia (IDA) | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Hb <10.5 g/dL during second trimester and Hb <11 g/dL during third trimester
Complete blood count (CBC) with differential (WBC, RBC, Hematocrit, MCV, MCH, MCHC, RDW, Platelet Count, MPV and Differential (Absolute and Percent - Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils) | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw
Maternal serum ferritin | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw
Maternal serum iron | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw
Maternal sTfR | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw
Maternal total body iron (TBI) | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  (TBI (mg/kg) = - [log(TfR/ferritin ratio) - 2.8229]/0.1207)
Maternal hepcidin | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw
Maternal erythropoietin (EPO) | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw
Maternal circulating cytokines (interleukin-6 (IL-6), GM-CS, IL-2, IL-4, IL-8, IL-10, TNFα, and IFNγ | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw
Maternal C-reactive protein (CRP) | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw
Maternal Erythroferrone (ERFE) | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Venous blood draw
Maternal Erythroferrone (ERFE) Cord Complete blood count (CBC) with differential (WBC, RBC, Hematocrit, MCV, MCH, MCHC, RDW, Platelet Count, MPV and Differential (Absolute and Percent - Neutrophils, Lymphocytes, Monocytes, Eosinophils, and Basophils) | delivery
  Cord blood draw
Cord serum ferritin | delivery
  Cord blood draw
Cord serum iron | delivery
  Cord blood draw
Cord sTfR | delivery
  Cord blood draw
Cord total body iron (TBI) | delivery
  (TBI (mg/kg) = - [log(TfR/ferritin ratio) - 2.8229]/0.1207)
Newborn heel stick | After delivery before baby released home
  Blood spot
Placenta iron transporter (FPN-1 and TFR-1) | delivery
  Western blot
Placenta iron quantification | delivery
  Immunohistochemistry
Placenta tissue iron concentration | delivery
  Inductively coupled plasma-mass spectrometry (ICP-MS)
Fecal abundance of A. muciniphila | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3), delivery (V4)
  Quantitative polymerase chain reaction (qPCR)
Shot-gun sequencing and analysis (taxonomy and functional profiling) | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3)
  MetaPhlAn4 and HUMAnN 2.0
Microbial mucin degrading enzymes | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3)
  CaZymes
Stool pH | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3)
  pH probe
Adverse pregnancy outcomes post-treatment and at delivery (clinical- EMR) | delivery
  Adverse pregnancy outcomes post-treatment and at delivery (clinical-EMR)
Probiotic acceptance and tolerability | 10-16 weeks GA, 14-20 weeks GA, 18-24 weeks GA, 22-28 weeks GA, 26-32 weeks GA, 30-36 weeks GA, 34-40 weeks GA, 38-40 weeks GA
  Daily capsule adherence Reported adverse health effects
Auditory Brainstem Response (ABR) testing | -3 days postpartum
  Interpeak latency I-V

OTHER OUTCOMES:
Habitual and recent dietary intake | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3)
  Food frequency (baseline only) questionnaire and 24-hour diet recall
Physical activity | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3)
  Self-report questionnaire
Infant characteristics (clinical-EMR) | delivery
  Infant sex, weight, gestational age (clinical-EMR)
Pre-pregnancy body mass index (BMI) | Up to 6 months before pregnancy
  Self-report (confirmed by clinical-EMR, if possible) BMI will be calculated as kg/m2
Gestational weight gain | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3)
  Gestational weight gain
Gut microbiome factors | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3)
  Questionnaire related to allergies, diet, travel, and environment
Presence of probiotic strain in stool | 10-16 weeks GA (V1), 22-28 weeks GA (V2), 30-36 weeks GA (V3)
  Quantitative polymerase chain reaction (qPCR)

IPD SHARING:
Plan to Share IPD: Undecided